CLINICAL TRIAL: NCT06001554
Title: Improving Adolescent Student Mental Health and Quality of Life Through a Reduction in Physical and Emotional Violence by Teachers in Pakistan: A Cluster Randomized Controlled Trial
Brief Title: Preventing Physical and Emotional Violence by Teachers in Public Schools in Pakistan
Acronym: ICC-T_Pak
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bielefeld University (Other)
Collaborators: Shifa Foundation (Unknown); Shifa International Hospital (Other); Mclean Hospital (Other); University of Konstanz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICC-T CRCT Pakistan
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-07

CONDITIONS: Violence
Keywords: school violence; teacher violence; teachers; intervention; students; public schools; secondary schools

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICC-T (Experimental): 5 days with 8 hours of training for teachers. Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Interventions: Behavioral: Interaction Competencies with Children - for Teachers (ICC-T)
- monitoring condition (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Interaction Competencies with Children - for Teachers (ICC-T) — Core training components include teacher-student interaction, maltreatment prevention, effective discipline strategies, identifying and supporting burdened students and implementation of the training materials into the school setting
  Arms: ICC-T

SUMMARY:
Violence has severe and long-lasting negative consequences for children and adolescents' well-being and psychosocial functioning, thereby also hampering communities and societies' economic growth. Studies show high prevalence rates of violence by teachers against children in Pakistan. In addition to legal and structural factors (e. g. stressful working conditions for teachers), attitudes favoring violence against children as an effective and acceptable discipline method and the lack of access to alternative non-violent strategies are likely to contribute to teachers' ongoing use of violence against children.

Notwithstanding, there are currently very few school-level interventions to reduce violence by teachers that a) have been scientifically evaluated and b) that focus both on changing attitudes towards violence and on equipping teachers with non-violent discipline strategies.

Thus, the present study tests the effectiveness of the preventative intervention Interaction Competencies with Children - for Teachers (ICC-T) in secondary schools in Pakistan. Previous studies have provided initial evidence on the feasibility to implement teacher violence interventions in secondary schools in Pakistan. This study aims to provide first evidence for the effectiveness of ICC-T to reduce violence and to improve children's functioning (i.e. mental health, well-being, academic performance) in Pakistan.

DETAILED DESCRIPTION:
The study is a multi-site cluster randomized controlled trial with schools (clusters) as level of randomization. Three districts in each site of the four sites (Khyber Pakhtunkhwa province, Sindh province, the State of Azad Jammu & Kashmir, and the federal capital Islamabad+Punjab province) will be purposely selected to ensure diversity of schools in terms of geographical, economical, social, and politically background. In each site, 12 public schools will be randomly selected, resulting in a total number of 48 schools (12 per sites). Schools will be stratified based on school type (girls or boys school). In each site, 6 schools (3 girls and 3 boys schools) will be randomly allocated to the intervention group (that will receive the ICC-T intervention) and the control group (that will receive no intervention).

At each school, 30 students in the first year of secondary and all teachers (expected average number: 15) will be recruited. Thus the final sample will comprise 1440 students and at least 720 teachers at baseline.

The study will have three data assessment points: baseline assessment prior to the intervention, the first follow-up assessment six months after the intervention and the second follow-up assessment 18 months after the intervention. In addition, feasibility data will be assessed in the intervention group at the beginning and the end of the intervention.

Primary outcome measures are student- and teacher-reported physical and emotional violence by teachers in the past week. Secondary outcome measures include children's emotional and behavioral problems, quality of life, cognitive functioning, academic performance, and school attendance.

ELIGIBILITY:
General:

Inclusion Criteria:

All: Written informed consent (if underaged by parents (written) & minors themselves (written) Students: Enrollment in selected secondary school Teachers: All teachers employed at the selected schools

Schools:

Public secondary schools Day schools At least 30 students in selected class/stream

Exclusion criteria:

Students and teachers:

Acute drug or alcohol intoxication Acute psychotic disorder

Ages: 11 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2100 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change of students' exposure to emotional and physical violence by teachers | The CTS will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess students' self-reported experiences of emotional and physical violence by teachers at school in the past week. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger reduction of exposure to violence in the intervention group compared to the control group.
Change of teachers' use of emotional and physical violence | The CTS will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  The Conflict Tactics Scale (CTS) will be used to assess teachers' use of emotional and physical violent discipline measures against students in the past week. Higher scores indicate higher levels of violence that is used by teachers. We hypothesize a stronger reduction of the use of violence in the intervention group compared to the control group.

SECONDARY OUTCOMES:
Change of teachers' positive attitudes towards emotional and physical violence | The adapted version of CTS will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after the intervention)
  Teacher's attitudes towards emotional and physical violence will be assessed with an adapted version of the Conflict Tactic Scale (CTS). Higher scores indicate higher levels of positive attitudes towards violence. We hypothesize a stronger decrease of positive attitudes towards violence in the intervention group compared to the control group.
Change of student's mental health | The PSC-Y will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  The Pediatric Symptom Checklist - Youth Report (PSC-Y) will assess students' emotional and behavioral problems.
  Higher scores indicate higher levels of students' mental health problems. We hypothesize a stronger reduction of mental health problems in the intervention group compared to the control group.
Change of students' quality of life | The KIDSCREEN-10 will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  The KIDSCREEN-10 will assess students' quality of life. Higher scores indicate higher levels of students' quality of life.
  We hypothesize an overall improvement of in the quality of life in the intervention group compared to the control group.
Change of students' cognitive functioning | The app-based tasks will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  Five tasks from the tablet application Inquisit will be used to assess children's cognitive abilities including selective attention (Letter Cancellation Task), working memory (Corsi Block Tapping Backwards), response inhibition (Arrow Flanker Task), planning and problem solving (Tower of London) and cognitive flexibility (Wisconsin Card Sorting Test). The test results in each test will be z-standardized and then combined to one compound score. Higher scores indicate higher levels of students' cognitive abilities. We hypothesize higher levels of cognitive functioning in the intervention group compared to the control group.

OTHER OUTCOMES:
Change of students' academic performance | Students' grades will be collected at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention).
  Students' grades in the previous term's exams will be obtained from the school administration. An improvement in academic performance in the intervention group is hypothesized.
Change of peer violence | he Multidimensional Peer Victimization Scale will be used at T0 (baseline, prior to intervention), T1 (first follow-up, 6 months after intervention) and T2 (second follow-up, 18 months after intervention)
  The Multidimensional Peer Victimization Scale will be used assess students' experiences of violence by peers. Higher scores indicate higher levels of students' experiences of peer violence. We hypothesize a stronger decrease of peer violence in the intervention group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Alaptagin Khan, MBBS, Principal Investigator — McLean Hopstial
Locations (1):
- Shifa International Hospitals, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The ICC-T intervention is being tested in various other countries including Haiti, Ghana, Tanzania and Uganda. We will share anonymized data with project partners from the different countries for combined and/or comparative analyses. In addition, we will share anonymized data with other researchers working on prevention of violence against children in school settings for the purpose of conducting synthesizing analyses such as meta-analyses.
  Finally, the anonymized data collected in the study will be made publicly available in a data repository.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The anonymized data will be made publicly available after completion of the project in 2027
Access Criteria: During the project, anonymized data will be shared only with partners working in other ICC-T projects and other researchers working in prevention of violence against children upon request. After the completion of the project, the anonymized data will be available to the public.

REFERENCES:
- [Derived] Khan A, Goessmann K, Scharpf F, Shah FKS, Kirika A, Azhar K, Yousafzai AW, Hoeffler A, Hecker T. Preventing physical and emotional violence by teachers in public schools in Pakistan: study protocol for a cluster-randomized controlled trial of the intervention Interaction Competencies with Children - for Teachers (ICC-T). BMC Public Health. 2025 May 24;25(1):1924. doi: 10.1186/s12889-025-23144-x. PMID 40413430